CLINICAL TRIAL: NCT00964327
Title: A Phase IIa Open-label, Randomized Trial to Determine the Antiviral Activity in 60 HIV Positive Subjects With Multiple PI Resistant Strains, Receiving Either Control Treatment or a Daily Dose of 800, 1600, 2400 or 3600 mg TMC114 (Darunavir) for 13 Days Followed by a Single Dose on Day 14
Brief Title: TMC114-C201: A Study to Determine the Antiviral Activity of TMC114 in Patients With Multiple Protease Inhibitor (PI) Resistant Human Immunodeficiency Virus (HIV) Strains
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals Limited, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006718
Record Dates: First submitted 2009-07-27; First posted 2009-08-24 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections
Keywords: TMC114-C201; TMC114; HIV; darunavir
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

INTERVENTIONS:
Drug: TMC114

SUMMARY:
The purpose of this study is to determine the antiviral activity, safety and tolerability of 14 days of different doses of TMC114 to treat HIV-1 positive patients whose condition is failing on a current treatment regimen that includes a protease inhibitor (PI) (a medication used to reduce the amount of HIV virus in the blood).To be considered for the study, patients must have a documented resistance to at least 2 of the current PIs. Pharmacokinetics and pharmacodynamics of TMC114 will also be assessed.

DETAILED DESCRIPTION:
This is a Phase lla open-label (all people involved know the identity of the treatment), randomized (study drug assigned by chance), controlled (the patients of the control group continue the failing regimen), dose-finding study to determine the antiviral activity, safety and tolerability of a 14-day treatment with TMC114 (a protease inhibitor) for treatment of human immunodeficiency virus type 1 (HIV-1) positive patients who are considered resistant to (failing to improve on) 2 or more protease inhibitors (PIs). Sixty HIV-1 positive patients, who are resistant to multiple PIs as confirmed by specialized testing (virtual phenotyping) and who are currently failing to improve on a treatment regimen that contains a PI, will be randomly assigned to one of 5 treatment groups. Those randomized to the control group will continue their current therapy (consisting of PIs and Nucleoside Reverse Transcriptase Inhibitor(s) (NRTIs)). Those randomized to the TMC114 treatment groups will receive the study drug as a substitute for all the PIs in the current failing treatment regimen at the following dose levels: 400 or 800 mg twice a day, or 800 or 1200 mg three times a day for 13 days followed by a single dose on day 14. The dose of the NRTIs (NRTIs are drugs that suppress replication of retroviruses) will remain unchanged until the end of the treatment period. The trial will involve a screening period of maximum three weeks, a 7-day run-in period (the period of time before study start when no treatment is given), a 14-day treatment period, followed by a 6- week follow-up period. The maximal trial duration will thus be twelve weeks. Primary objective is to determine the antiviral activity of TMC114 as well as the pharmacokinetics (how the drug is absorbed in the body, distributed within the body and how it is removed from the body over time) and pharmacodynamics (the study of the action of effects a drug has on the body) will also be assessed over the 2 week period.Safety will be followed at regular intervals during treatment and follow-up period. Safety assessments consist of regular lab assessments, ECG recording, vital signs, physical examination, body weight and Body Mass Index. Observation of and interview for adverse events will be done daily during the first week of treatment, every second day during the 2nd week of treatment, and at week 1, 3 and 6 of the follow-up period. In addition an Independent Data Monitoring Committee will evaluate the study data at regular intervals. Patients will be randomly assigned to one of 5 treatment groups: 400 or 800 mg twice a day for 13 days followed by a single dose on day 14, or 800 or 1200 mg three times a day for 13 days followed by a single dose on day 14. Patients randomized to the control group will continue their current therapy consisting of protease inhibitors (PIs) and Nucleoside Reverse Transcriptase Inhibitors (NRTIs).

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented HIV-1 infection with a viral load at screening visit above 2,000 HIV copies/ml
* Currently treated with a failing antiretroviral regimen consisting of NRTIs together with one or more PI(s)
* Has a resistance against at least 2 of the currently used PIs
* Patient agrees not to change the current therapy until end of run-in and agrees not to change NRTIs until the end of treatment period
* No current AIDS defining illnesses

Exclusion Criteria:

* NNRTI (non-nucleoside reverse transcriptase inhibitor) containing regimen, two weeks prior to screening
* Suspicion of alcohol abuse or drug abuse, leading to non-compliance
* History of significant drug allergy induced by PIs
* CD4 count < 50
* Life expectancy of less than 6 months
* Pregnant or breast feeding females
* Females of childbearing potential without use of a highly effective birth control method or not willing to continue practicing this birth control method for at least 14 days after the end of the treatment
* Received an investigational drug within 30 days prior to the trial drug administration
* Patients with clinically significant laboratory abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-08; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To determine the antiviral activity of TMC114. | Screening, days -7, -3, 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14 , 15, follow-up weeks 1, 3 and 6

SECONDARY OUTCOMES:
nadir of viral load | Screening, days -7, -3, 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14 , 15, follow-up weeks 1, 3 and 6
Pharmacokinetics (PK) / Pharmacodynamics (PD): Plasma concentration of TMC114 and efficacy and safety data will be analyzed to find relationships between PK and PD. | 12 visits
CD4 count | 7 visits

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Clinical Study Report Synopsis of TMC114-C201: A study to determine the antiviral activity of TMC114 in patients with multiple protease inhibitor (PI) resistant human immunodeficiency virus (HIV) strains. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=991&filename=CR006718_CSR.pdf